CLINICAL TRIAL: NCT06173050
Title: Internal Evaluation of PAP Systems: Comparison of PAP Flow Generators Machines, Mask Systems and Tubing
Brief Title: PAP Systems Internal Clinical Studies (ICS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SLP-23-10-01
Record Dates: First submitted 2023-11-09; First posted 2023-12-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: This is an open label, prospective, randomized cross over (or single arm) study designed to support the development of new accessories for PAP devices.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAP System A (with Amalfi) then PAP System B (with CLA11) (Other): Participants will be asked to take home the investigational PAP system (Amalfi) to use at night while they sleep in place of their own PAP system. The participant's therapy and comfort settings will not be altered. Participants will be randomized as to the order they will trial PAP System A and PAP System B. This arm will first use the Amalfi for 7 days and then use the CLA 11 for 7 days.
  Interventions: Device: PAP System A (with Amalfi) then PAP System B (with CLA11)
- PAP System B (with CLA11) then PAP System A (with Amalfi) (Active Comparator): Participants will be asked to take home the comparator PAP system B (CLA 11) to use at night while they sleep in place of their own PAP system. The participant's therapy and comfort settings will not be altered. Participants will be randomized as to the order they will trial PAP System B and PAP System A. This arm will first use the CLA 11 for 7 days and then use the Amalfi for 7 days.
  Interventions: Device: PAP System B (with CLA11) then PAP System A (with Amalfi)

INTERVENTIONS:
Device: PAP System A (with Amalfi) then PAP System B (with CLA11) — PAP System A (with Amalfi) for 7 days followed by PAP System B (with CLA11) for 7 days
  Arms: PAP System A (with Amalfi) then PAP System B (with CLA11)
Device: PAP System B (with CLA11) then PAP System A (with Amalfi) — PAP System B (with CLA11) for 7 days followed by PAP System A (with Amalfi) for 7 days
  Arms: PAP System B (with CLA11) then PAP System A (with Amalfi)

SUMMARY:
This is a pre-market study for ongoing product development aiming to explore the usability and performance of the study PAP systems to guide product development.

DETAILED DESCRIPTION:
This is an open label, prospective, randomized cross over (or single arm) study designed to support the development of new accessories for PAP devices. This generic protocol provides a framework methodology for how these ongoing studies will be conducted. This protocol then is used in a number of smaller sub-studies, each of which will have their own sub-protocol outlining the exact specifics of the study.

The studies could be run face-to-face or remotely.

Participants are healthy volunteers who are ResMed employees. Recruitment will be done via emails. Participants will be explained the details of the trial and those who wish to take part will be invited to a selected site for the first study visit.

Visit 1: Participants will provide written informed consent. Participants will be shown the PAP systems and trial them for fit and comfort. Participants may be asked initial questions on their first thoughts on the PAP systems. If the participant and assessor are happy to proceed, the participants will use the loan PAP system for trial.

Visit 2: After trialing the PAP systems, participants will be asked to complete a questionnaire regarding the appeal, comfort, and usability of the PAP system(s). Depending on sub-study protocol, participants will then take the second PAP system home to test.

Visit 3: The participant will return the loan PAP system to the assessor. The participants' questionnaire responses will be reviewed. This concludes the participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are employees of ResMed
* Participants shall be volunteers
* Participants willing to give written informed consent
* Participants who ≥ 18 years of age
* Participants willing and able to complete the specified tasks

Exclusion Criteria:

* Participants who are or may be pregnant.
* Participants with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Participants believed to be unsuitable for inclusion by the researcher.
* Participants who or whose bed partner has implantable medical devices which may contraindicate against masks with magnetic clips (exclusion criteria for study masks with magnetic clips only)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Subjective outcomes parameters scores | 6 weeks
  Subjective outcomes parameters scores from participants. Each subjective outcomes item of the investigational component/s of the PAP System will be rated on a Likert Scale questionnaire. Scores will be collected using an 11-point Likert Scale Questionnaire. Minimum value will be zero. Maximum value will be 10. A higher score indicates better outcomes. A score of 10 is considered very favorable, and a score of 0 is very unfavorable.

IPD SHARING:
Plan to Share IPD: No